CLINICAL TRIAL: NCT06359561
Title: Assessment of Effectiveness and Stimulation Coverage of Closed-loop Spinal Cord
Brief Title: Assessment of Effectiveness and Stimulation Coverage of Closed-loop Spinal Cord Stimulation (CL-SCS) Therapy in Patients with Cervical Lead Placement
Status: Enrolling by invitation | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Collaborators: Saluda Medical Pty Ltd (Industry)
Responsible Party: Principal Investigator, Jan Willem Kallewaard phd, MD PhD dr., Rijnstate Hospital
Other Study IDs: 2023-2201 - Cervical lead
Record Dates: First submitted 2024-02-27; First posted 2024-04-11 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pain Syndrome; Multi Focal Pain; Failed Neck Surgery Syndrome; Polyneuropathies
Keywords: Spinal cord stimulation; Cervical lead placement; Closed loop stimulation; Multi focal pain
MeSH Terms: conditions — Polyneuropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- single arm: Up to 40 subjects eligible for SCS trial and permanent implant with a minimum of pain intensity of 5/10 on NRS at baseline will be enrolled.
  Interventions: Device: cervical lead placement

INTERVENTIONS:
Device: cervical lead placement — implant of cervical lead neurostimulation, using saluda medical devices

SUMMARY:
This observational, prospective data collection is designed to evaluate the effectiveness and stimulation coverage of closed-loop spinal cord stimulation (CL-SCS) therapy in patients with cervical lead placement.

DETAILED DESCRIPTION:
Title Assessment of effectiveness and stimulation coverage of closed-loop spinal cord stimulation (CL-SCS) therapy in patients with cervical lead placement.

Device used in the study The Saluda Medical EvokeTM Closed-Loop Spinal Cord Stimulator (CL-SCS) System (Evoke System). The CE marked Evoke System will be used within its licensed use and manuals. The Evoke System measures and records spinal cord (SC) activation resulting from stimulation via evoked compound action potentials (ECAPs). The Evoke System can be programmed to provide ECAP-controlled, closed-loop SCS or open-loop, fixed-output (traditional) SCS; ECAPs may be measured and recorded in either stimulation mode.

Indication for use The Evoke SCS System is indicated as an aid in the management of chronic intractable pain of the trunk and/or limbs and will be used within its licensed indication during this study.

Rational This observational, prospective data collection is designed to evaluate the effectiveness and stimulation coverage of closed-loop spinal cord stimulation (CL-SCS) therapy in patients with cervical lead placement.

Study design An observational, prospective, multi-center, single-arm study. Study population Up to 40 subjects eligible for SCS trial and permanent implant with a minimum of pain intensity of 5/10 on NRS at baseline will be enrolled.

Objectives

* Evaluate stimulation coverage in pain area and other parts of the body, sensation (awareness and quality) and pain relief using a 0-10 numeric rating score (NRS) in patient implanted with one or two leads at cervical level receiving closed-loop spinal cord stimulator (CL-SCS) therapy.
* Assessment of holistic outcomes: measure quality of life in seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) assessed by the PROMIS-29 questionnaire.
* Evaluate medication intake, patient satisfaction and patient global impression of change (PGIC).
* Assessment of device data and programming parameters.
* Neurophysiological measurements: neuronal activation, conduction velocity and posture change assessment.

Inclusion criteria

* Subject is deemed a suitable candidate for SCS trail and permanent implant and has been routinely scheduled to undergo an SCS trial phase with the Evoke SCS System.
* Subject is ≥ 18 years old.
* Subject is not pregnant or nursing.
* Subject is willing and capable of giving informed consent. Exclusion criteria
* Subject currently has an active implantable device including pacemakers, spinal cord stimulator or intrathecal drug delivery system.
* Subject is incapable of understanding or responding to the study questionnaires.
* Subject is incapable of understanding or operating the patient programmer handset.

Burden and Risk

* There will be no additional burden associated with participation in the study. The data will be collected during the standard of care visits. Data collection required by the study protocol will add no additional time to standard clinical appointments, as the data will be downloaded from the clinical interface or entered directly into the database.
* The benefits of this study could enable improved treatment of chronic trunk and/or limb pain with the closed loop system and cervical lead placement.

ELIGIBILITY:
Inclusion Criteria:

* Subject is deemed a suitable candidate for SCS trail and permanent implant and has been routinely scheduled to undergo an SCS trial phase with the Evoke SCS System.
* Subject is ≥ 18 years old.
* Subject is not pregnant or nursing.
* Subject is willing and capable of giving informed consent.

Exclusion Criteria:

* Subject currently has an active implantable device including pacemakers, spinal cord stimulator or intrathecal drug delivery system.
* Subject is incapable of understanding or responding to the study questionnaires.
* Subject is incapable of understanding or operating the patient programmer handset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for SCS trial and permanent implant will be recruited to participate in the study. Subjects will read and sign an informed consent prior to study participation. Subjects meeting all the inclusion and none of the exclusion criteria and receiving a permanent implant with cervical lead placement will be considered enrolled. Up to 40 subjects receiving a permanent implant will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity in pain region(s) of pain using the 11-box pain numeric rating scale (NRS) | baseline, 3months, 6 months, 12 months
  NRS scoring: 0 no pain, 10 worst imaginable pain

SECONDARY OUTCOMES:
Pain distribution using Patient Reported Dermatomal Coverage Map | baseline, 3months, 6 months, 12 months
  Subjects will be asked to map and track pain distribution (extent and location) by shading in the areas where they typically experience pain on a body map drawing. "Shade in the areas where you typically experience "study pain" on the pain map below. If the pain goes from front to back, then shade in those areas on each side of the picture."
Assessment of holistic outcomes: quality of life in seven domains (physical function, fatigue, pain interference, depression, anxiety, ability to participate in social roles and activities, and sleep disturbance) assessed by the PROMIS-29 questionnaire | baseline, 3months, 6 months, 12 months
  The PROMIS 29+2 Profile v2.1 is a 29-item profile instrument that assesses 8 universal domains (not disease-specific): Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles and Activities, Pain Interference, and Pain Intensity. The first seven domains are assessed with 4 questions each. High scores represent more of the domain being measured. Thus, on symptom-oriented (negatively worded) domains of PROMIS 29+2 Profile v2.1 (anxiety, depression, fatigue, pain interference, and sleep disturbance), higher scores represent worse symptomatology. On the function-oriented (positively worded) domains (physical functioning and social role) higher scores represent better functioning. Pain Intensity is measured with a single 11-point numeric rating scale (NRS) from 0 (no pain) to 10 (worst imaginable pain).
Pain-related medication intake. | baseline, 3months, 6 months, 12 months
Programming parameters. | 3months, 6 months, 12 months
  Program parameters (e.g., leads programmed: configuration ) will be collected. This data is automatically recorded on the SCS-device.
Programming parameters. | 3months, 6 months, 12 months
  Program parameters (e.g., pulsed width recorded in unit: micro seconds) will be collected. This data is automatically recorded on the SCS-device.
Evaluate stimulation sensation (awareness and quality) | 3months, 6 months, 12 months
  Subject will be asked how aware he/she is of the stimulation sensation and is presented with a 5-point rating scale containing the options "Always aware of stimulation sensation", "Usually aware of stimulation sensation", "Sometimes aware of stimulation sensation", "Rarely aware of stimulation sensation", and "Never aware of stimulation sensation". Subjects will be asked a question about stimulation sensation quality and can rate from "Unpleasant", "Neither pleasant nor unpleasant", "Pleasant" to "No sensation".
Evaluate stimulation coverage in pain region(s) | 3months, 6 months, 12 months
  Subjects will be asked to map and track stimulation distribution (extent and location) by shading in the areas where they typically experience stimulation sensation on a body map drawing. "Shade in the areas where you typically experience stimulation on the body map below. If the stimulation goes from front to back, then shade in those areas on each side of the picture."
Posture Change Measurements | 6 months, 12 months
  Data on stimulation intensity and ECAP amplitude at various stimulation levels (i.e., activation plot) and in different postures will be collected in both stimulation modes. Subjects will rate the stimulation intensity on an 11-point numeric rating scale (0 equals "no feeling" and 10 equals "very intense"). All these measurements are automatically recorded on the device except subject ratings, which will be recorded on the CRF.

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] Cameron T. Safety and efficacy of spinal cord stimulation for the treatment of chronic pain: a 20-year literature review. J Neurosurg. 2004 Mar;100(3 Suppl Spine):254-67. doi: 10.3171/spi.2004.100.3.0254. PMID 15029914
- [Background] Deer TR, Mekhail N, Provenzano D, Pope J, Krames E, Leong M, Levy RM, Abejon D, Buchser E, Burton A, Buvanendran A, Candido K, Caraway D, Cousins M, DeJongste M, Diwan S, Eldabe S, Gatzinsky K, Foreman RD, Hayek S, Kim P, Kinfe T, Kloth D, Kumar K, Rizvi S, Lad SP, Liem L, Linderoth B, Mackey S, McDowell G, McRoberts P, Poree L, Prager J, Raso L, Rauck R, Russo M, Simpson B, Slavin K, Staats P, Stanton-Hicks M, Verrills P, Wellington J, Williams K, North R; Neuromodulation Appropriateness Consensus Committee. The appropriate use of neurostimulation of the spinal cord and peripheral nervous system for the treatment of chronic pain and ischemic diseases: the Neuromodulation Appropriateness Consensus Committee. Neuromodulation. 2014 Aug;17(6):515-50; discussion 550. doi: 10.1111/ner.12208. PMID 25112889
- [Background] Turner JA, Loeser JD, Deyo RA, Sanders SB. Spinal cord stimulation for patients with failed back surgery syndrome or complex regional pain syndrome: a systematic review of effectiveness and complications. Pain. 2004 Mar;108(1-2):137-47. doi: 10.1016/j.pain.2003.12.016. PMID 15109517
- [Background] Surges G, Paulus J, Blass T, Mendryscha K, Bettag M, Rotte A. Efficacy and Safety of 10 kHz Spinal Cord Stimulation Using Cervical and Thoracic Leads: A Single-Center Retrospective Experience. Pain Ther. 2021 Dec;10(2):1255-1268. doi: 10.1007/s40122-021-00287-4. Epub 2021 Jul 8. PMID 34236671